CLINICAL TRIAL: NCT02937688
Title: Deep Brain Stimulation (DBS) for Parkinson's Disease International Study (REACH-PD)
Brief Title: Deep Brain Stimulation (DBS) for Parkinson's Disease International Study
Acronym: REACH-PD
Status: Completed | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Other Study IDs: 1678
Record Dates: First submitted 2016-10-17; First posted 2016-10-18 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Medtronic DBS Therapy for Parkinson's disease — Bilateral Deep Brain Stimulation (DBS) of the Subthalamic Nucleus or Globus Pallidus interna.
  Other Names: Medtronic Activa DBS System

SUMMARY:
To gather data on DBS Therapy effectiveness in different geographic populations.

DETAILED DESCRIPTION:
The purpose of this prospective open label post market study of DBS for PD is to gather data on DBS therapy effectiveness as measured by clinician and patient reported health outcomes data through one year of follow-up in different geographic populations.

ELIGIBILITY:
Inclusion Criteria:

1. Indication of DBS for PD consistent with the country specific approved labeling.
2. Levodopa-responsive Parkinson's disease (UPDRS III ≥ 30% improvement on Levodopa challenge test).
3. Symptoms treatable by medications but not adequately controlled with medications (with persistent disabling symptoms, such as motor fluctuations, dyskinesia).
4. At least 22 years old.
5. Screening cranial MRI, performed within 12 months of entry into the study, that is normal or with a non-significant abnormality that does not present any incremental risks or concerns for the patient as a result of the DBS procedure.
6. Understand potential risk/benefit, consent to the study, study procedures, and agree to complete the study follow-up visits and comply with the study protocol requirements.

Exclusion Criteria:

1. Secondary Parkinson's disease, atypical syndromes.
2. Previous stereotactic functional neurosurgery or ablative therapy (e.g., pallidotomy, subthalamotomy), surgical contraindications related to DBS.
3. Dementia (Mattis Dementia Rating Scale ≤ 130), major depression with suicidal thoughts (Beck Depression Inventory II > 25), acute psychosis, active alcohol or drug abuse, terminal illness, and any major medical or psychological histories, diagnoses, conditions, or comorbidities that would interfere with participation in the study per the investigator's medical judgment.
4. Electrical or electromagnetic implant (e.g., Cochlear prosthesis, cardiac pacemaker).
5. Surgical or medical contraindications to DBS surgery or therapy (e.g., uncontrolled hypertension, advanced coronary artery disease).
6. Participation in a drug, device, or biologics trial within the preceding 30 days that may confound the study results.
7. Pregnant female.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with levodopa responsive Parkinson's disease that are not adequately controlled by medication.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Parkinson's disease-related quality of life, as measured by the Parkinson's Disease Questionnaire (PDQ-8). | Baseline to 12 months
Change in motor score, as measured by the Unified Parkinson's Disease Rating Scale (UPDRS) III, off medication | Baseline to 12 months

CONTACTS AND LOCATIONS:
Locations (15):
- Brazil (8):
  - Hospital Universitário Cajuru, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Hospital Sao Rafael - Monte Tabor, Salvador
  - Hospital de Base de São Jose do Rio Preto, São José do Rio Preto
  - Hospital das Clinicas de Sao Paulo/ IPQ, São Paulo
  - SPDM- Hospital Sao Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo
- China (7):
  - Xuanwu Hospital Capital Medical University, Beijing
  - Huaxi Hospital, Chengdu
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - Huashan Hospital, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - Tangdu Hospital, Xi'an

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Chen L, Sun B, Wang X, Wang J, Wang J, Woods J, Stromberg K, Shang H. Quality of Life and Motor Outcomes in Patients With Parkinson's Disease 12 Months After Deep Brain Stimulation in China. Neuromodulation. 2023 Feb;26(2):443-450. doi: 10.1016/j.neurom.2022.10.047. Epub 2022 Nov 18. PMID 36411150